CLINICAL TRIAL: NCT04266873
Title: Measurement of Mucus Plugging With Computer Tomography Before and Following Implementation of the AffloVest in Adults With Bronchiectasis - a Feasibility Study'
Brief Title: Feasibility Study of the AffloVest in Bronchiectasis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Data analysis review of current data
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO2552
Record Dates: First submitted 2020-01-13; First posted 2020-02-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Feasibility interventional study using intervention for 6 weeks
Masking Description: CT scans will be anonymised before being sent to Radiographer to Brody score
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AffloVest HFCWO intervention (Experimental): Use of the AffloVest for 30 mins, twice a day for 6 weeks
  Interventions: Device: AffloVest

INTERVENTIONS:
Device: AffloVest — Form of High Frequency Chest Wall Oscillation mimicking manual techniques on a patients thorax to assist with secretion clearance. Delivered for 30 minutes, twice a day

SUMMARY:
Feasibility study of High Frequency Chest Wall Oscillation (HFCWO) using the AffloVest in 30 patients with Bronchiectasis over a 6 week period. Outcome measures include lung function, quality of life questionnaire, High resolution computed Tomography and visual analogue scale for ease of clearance.

DETAILED DESCRIPTION:
The study is an feasibility study evaluating the impact of using the AffloVest for 30 minutes twice daily [in addition to their standard airway clearance regimen] for 6 weeks.

The study will endeavour to recruit 30 adult subjects (male and female) who have a known diagnosis of bronchiectasis and who attend the Cambridge Centre for Lung Infection (CCLI) at the Royal Papworth Hospital, Cambridge, United Kingdom.

Bronchiectasis is defined as symptoms of chronic or recurrent bronchial infection with radiological evidence of abnormal and permanent dilation of bronchi, not from cystic fibrosis. Subjects will be recruited through convenience sampling and must demonstrate stability during a 2-week period prior to enrolment. Stability is defined as no change in medical treatment.

Participants will use the AffloVest for 30 minutes twice dally [in addition to their standard airway clearance regimen] for 6 weeks (days 0 - 42). Clinical review and a serial testing will be completed at day1, day 21 and day 42 (at commencement of intervention, after 3 weeks intervention and after 6 weeks intervention) including high resolution computer tomography (HRCT) at full inspiration and full expiration; spirometry (FEV1 and FVC); and the patient reported outcomes Visual Analogue Scale for ease of sputum clearance (VAS), St George's Respiratory Questionnaire (SGRQ) and Quality of Life -Bronchiectasis (QOL-B).

HRCT imaging will be done at full inspiration and full expiration and scored by two independent expert thoracic radiologists using the validated Brody Scoring System which is sensitive and reproducible.

Both will be blinded to the timepoint of the HRCT being analysed and if there is disagreement in scores an average will be taken.

We hypothesize that changes in HRCT score and patient reported outcomes will be seen post treatment with the AffloVest, confirming it as an efficacious therapy for airway clearance in adults with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and females 18 years or over
* Current diagnosis of bronchiectasis
* Productive of sputum on a daily basis
* Clinical stability over a 2 week period prior to enrolment

Exclusion Criteria:

* Cystic fibrosis
* Severe obstructive airways disease (defined as FEV1 less than 25 percent)
* Predominant lung disease is not bronchiectasis in the opinion of the investigator (e.g. asthma, Chronic Obstructive Pulmonary Disease (COPD), pulmonary fibrosis)
* Bronchiectasis in only 1 lobe
* Currently treated non-tuberculous mycobacterial lung disease
* Acute congestive cardiac failure
* Contra-indication or unable to perform HRCT imaging, including pregnancy
* Contra-indication to using AffloVest including lung malignancy, recent rib fractures, radiological evidence of lung cavitation, and recent significant haemoptysis (in the opinion of the investigator)
* History of poor adherence to physiotherapy treatment
* Cognitive or memory problems affecting ability to follow instructions or give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
High Resolution Computed Tomography (HRCT) | 6 weeks
  HRCT will be done at full inspiration and full expiration and reviewed by two independent radiographers who will be blinded to timepoint and participant. Radiographers will then use the Brody score to give the scans a score reflecting any changes to sputum volume or otherwise from intervention. Scans will be done and reviewed at baseline, three weeks of intervention and six weeks of intervention

SECONDARY OUTCOMES:
Forced Expiratory Volume at 1 second (FEV1) | 6 weeks
  FEV1, the forced air expelled at 1 second will be measured at baseline, after three weeks intervention and after six weeks intervention
Visual Analogue Score for ease of sputum expectoration (VAS) | 6 weeks
  A likert scale from 0-10 will be used for participants to score how easy it is for them to expectorate. Again, this will be assessed at baseline, after 3 weeks intervention and after 6 weeks intervention. 0 will be very easy to clear and 10 will be very difficult to clear
Quality of Life in Bronchiectasis questionnaire (QOL-B) | 6 weeks
  This subjective questionnaire will be completed as baseline, after three weeks intervention and after six weeks intervention. This is completed by the patient to assess how symptoms affect the quality of their lives. Final scores will be between 0 and 100 with higher scores representing better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Papworth Hospital NHS Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All participant specific data will be anonymised before any data will be published or shared

DOCUMENTS (2):
  • Study Protocol (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04266873/Prot_000.pdf
  • Informed Consent Form (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT04266873/ICF_001.pdf